CLINICAL TRIAL: NCT04905069
Title: Effectiveness of the SpaceOAR Vue System in Subjects With Prostate Cancer Being Treated With Stereotactic Body Radiotherapy
Acronym: SABRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U0702
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Stereotactic Body Radiotherapy; SBRT; Spacer; SpaceOAR; SpaceOAR Vue; Hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- No-Spacer Control (No Intervention): Subjects will receive radiotherapy without the use of the SpaceOAR Vue.
- SpaceOAR Vue (Experimental): Subjects will receive radiotherapy following injection of the SpaceOAR Vue hydrogel.
  Interventions: Device: SpaceOAR Vue System

INTERVENTIONS:
Device: SpaceOAR Vue System — The SpaceOAR Vue System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of the SpaceOAR Vue System to reduce the radiation dose delivered to the anterior rectum.
  The SpaceOAR Vue System is composed of biodegradable material, maintains space for the entire course of prostate radiotherapy treatment and is completely absorbed by the patient's body over time.
  Arms: SpaceOAR Vue

SUMMARY:
To demonstrate the effectiveness of the SpaceOAR Vue System in reducing late gastrointestinal (GI) toxicity in subjects undergoing Stereotactic Body Radiotherapy (SBRT) to treat prostate cancer.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of the SpaceOAR Vue System in reducing late gastrointestinal (GI) toxicity in participants undergoing Stereotactic Body Radiotherapy (SBRT) for the treatment of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Subjects must have pathologically confirmed (by routine hematoxylin and eosin (H&E) staining) invasive adenocarcinoma of the prostate and been planning to undergo SBRT.
* Subjects must have intermediate risk prostate cancer as defined by the presence of one or more of the following:
* Clinical Stage T2b - T2c (AJCC 6th edition) tumor
* Gleason Score 7 as determined from a biopsy taken within 9 months preceding Enrollment (randomization)
* Demonstrated blood PSA levels 10-20 ng/ml as measured within 6 months preceding Enrollment (randomization) and prior to commencing androgen deprivation therapy (ADT)
* Subject or authorized representative was informed of the nature of the study and provided written informed consent, approved by the appropriate Institutional Review Board (IRB)/Ethics Committee (EC) of the respective clinical site.

Exclusion Criteria:

* Prostate >80 cc documented within 9 months preceding Enrollment (randomization)
* Clinical stage T3 or T4 (AJCC 6th edition) tumor
* Blood PSA level >20 ng/ml as measured within 6 months preceding Enrollment (randomization) and prior to commencing androgen deprivation therapy (ADT)
* Gleason Score ≥ 8 as determined from a biopsy taken within 9 months preceding Enrollment (randomization)
* Subjects who had MRI evidence of gross posterior extracapsular extension (ECE) of the prostate cancer. (Note: MRI should be from within 9 months preceding Enrollment (randomization). If MRI is contraindicated, a digital rectal exam may be performed to confirm the absence of gross posterior ECE)
* Subjects who had metastatic disease, other ongoing cancers which were treated during the study or subjects for whom pelvic lymph node radiotherapy was planned.
* Subjects with any prior invasive malignancy (except non-melanomatous skin cancer) unless the subject had been disease free for a minimum of 3 years.
* History of prostatectomy, transurethral prostate surgery (e.g. TUNA, TUMT, TURP) if performed within 1 year prior to screening, other local prostate cancer therapy (e.g., cryotherapy or brachytherapy) or previous pelvic irradiation at any time prior to screening.
* History of prior pelvic surgery requiring low anterior or abdominoperineal resections or rectal surgery.
* History of or active inflammatory bowel disease (IBD) such as Crohn's disease or ulcerative colitis.
* History of or current perirectal disease that may interfere with interpretation of study outcomes including anal or perianal diseases such as fistula.
* Bleeding hemorrhoids requiring medical intervention within the prior three months.
* Diagnosed active bleeding disorder or a clinically significant coagulopathy. Note: Patients on anticoagulants may be included if the anticoagulant medication can be discontinued for index procedure.
* Active inflammatory or infectious process involving the perineum, gastrointestinal (GI) or urinary tract based on positive diagnosis or suspected diagnosis in the presence of fever >38⁰ C, WBC > 12,000/uL.
* Compromised immune system or prior diagnoses for human immunodeficiency virus (HIV) (with a detectable viral load within the last 6 months)/acquired immunodeficiency syndrome (AIDS) or autoimmune disease.
* If a subject was enrolled in another investigational drug or device trial that had not completed the primary endpoint or that clinically interfered with this study.
* Unable to comply with the study requirements or follow-up schedule.
* Any condition the Investigator believed would interfere with the intent of the study or would make participation not in the best interest of the patient.
* Known iodine sensitivity or allergy
* Known polyethylene glycol (PEG) sensitivity or allergy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Late Gastrointestinal (GI) Toxicity | 3 to 24 months post-SBRT initiation
  Proportion of subjects experiencing late GI toxicity after SBRT treatment with or without placement of the SpaceOAR Vue System hydrogel. Late GI toxicity is defined as the occurrence of a Grade 2 or greater GI adverse event (NCI CTCAE v4) between 3- and 24-months post-SBRT initiation

SECONDARY OUTCOMES:
EPIC-26 bowel score | 24 months post-SBRT initiation
  Proportion of subjects experiencing a decrease in EPIC-26 bowel score greater than or equal to the minimal important difference (MID) in EPIC-26 bowel score from baseline to 24 months post-SBRT initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Suneil Jain, MB, BCh, PhD, Principal Investigator — Queen's University, Belfast
Locations (30):
- United States (7):
  - GenesisCare USA, Fort Myers, Florida
  - Florida Urology Partners, LLC, Tampa, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - GenesisCare USA, Troy, Michigan
  - New Jersey Urology, a Summit Health Company, Bloomfield, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dr. John Sylvester, Myrtle Beach, South Carolina
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Princess Alexandra Hospital - ROPAIR, Woolloongabba, Queensland
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- France (2):
  - Institut Gustave Roussy, Villejuif, Cedex
  - Institut de Radiothérapie & Radiochirurgie HARTMANN, Levallois-Perret
- Germany (2):
  - MEDICLIN Robert Janker Klinik, Bonn
  - Klinikum Nurnberg Nord, Nuremberg
- Bon Secours Radiotherapy Cork, Cork, Ireland
- Italy (3):
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Policlinico Universitario Agostino Gemelli, Rome
  - IRCCS Ospedale Sacro Cuore Don Calabria, Verona
- Spain (3):
  - Hospital Universitario Cruces, Barakaldo
  - GenesisCare, Hospital San Francisco de Asis, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- Switzerland (2):
  - University Hospital Basel, Basel
  - Inselspital - University Hospital Bern, Bern
- United Kingdom (7):
  - Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey
  - Velindre Cancer Centre, Cardiff, Wales
  - Belfast City Hospital, Belfast
  - Bristol Haematology and Oncology Centre, Bristol
  - Royal Marsden Hospital, London
  - Norfolk and Norwich University Hospital NHS Trust, Norwich
  - Derriford General Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No